CLINICAL TRIAL: NCT04822857
Title: The Impact of Menopause on the Development of Heart Failure and Organ Damage of Hypertension
Status: Completed | Type: Observational
Sponsor: Polish Mother Memorial Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Kamil Janikowski, Medical Doctor, Polish Mother Memorial Hospital Research Institute
Other Study IDs: PolishMMHRI-BCO.5/2019
Record Dates: First submitted 2021-03-24; First posted 2021-03-30 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Hypertension; Menopause
Keywords: menopause; hypertension; estradiol; organ damage
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: AMH > cut-off point
  Interventions: Diagnostic Test: AMH
- 2: AMH < cut-off point
  Interventions: Diagnostic Test: AMH

INTERVENTIONS:
Diagnostic Test: AMH — The group was divided according to the level of Anti-Müllerian Hormone

SUMMARY:
Introduction: The average age of menopause in the Polish population is around 50 years. After the occurrence of the last menstruation in the woman's body there are series of hormonal changes that may result in the emergence of new diseases, i.e. osteoporosis or ischemic heart disease. Hypertension is the most important cardiovascular risk factor affecting morbidity and mortality due to cardiovascular disease. It is estimated that there are as many as 34% of adult Poles. The incidence of hypertension increases with age in both women and men, and significantly greater increases are observed in perimenopausal women. An equally important and growing health and economic problem in Poland is heart failure. It is estimated that up to 700,000 patients in our country are struggling with this disease, and the proportion of women in this group is constantly growing. This is the third reason for the death of women in Poland, causing more deaths than cancer. The influence of menopause on the occurrence of heart failure in a group of women with controlled hypertension remains unclear and is the subject of ongoing research. Similarly, there is still no convincing data on the increased risk of organ complications of arterial hypertension in the group of postmenopausal women.

The aim of the study is to assess the effect of menopause on myocardial function indexes, haemodynamic parameters and body mass composition in women aged> 40 years.

Material: about 100 women hospitalized in the Department of Cardiology and Congenital Heart Diseases of Adults > 40 years of age will be enrolled in the study. with controlled hypertension. The population will be divided into two groups: I: 50 women before the onset of menopause and II group: 50 women ≥ 1 year after the onset of menopause.

Methods: Basic laboratory tests and concentrations of ADMA, NT-proBNP, neprilysin, estradiol and FSH will be performed in patients. The other planned examinations are: full clinical examination with BMI assessment, resting ECG test, full echocardiography using tissue doppler, volume and function of the left atrium and vascular stiffness index assessed using the sphygmocor device. In addition, it is planned to analyze the composition of body mass using electrical bioimpedance, intima-media complex measurement and spiroergometric study. One year after the inclusion in the study, a telephone interview will be carried out with the patients, with particular attention to the diagnosed diseases / onset of intervention: heart failure, diabetes, atrial fibrillation, the need for coronary angiography or rehospitalisation. The collected data will be statistically processed.

New values: Studies carried out as part of this work will supplement the current knowledge on the impact of menopause in the population of women with hypertension on the risk of heart failure and complications of organ hypertension. Thanks to the observed relationships, it will be possible to early start the appropriate diagnostic procedure, the selection of personalized treatment and the development of a model of cardiac care for women in the perimenopausal period, and thus improve quality and extend their life.

DETAILED DESCRIPTION:
Introduction:

The average age of menopause in the Polish population is around 50 years. After the last menstruation a number of hormonal changes occur in the female body: estrogen, ovarian androgens (testosterone, androstenedione) and adrenal ones (DHEA, DHEAS), progesterone, growth hormone and insulin-like growth factors decrease. The concentration of gonadotropins gradually increases. These hormonal changes may result in the appearance of osteoporosis, climacteric syndrome, depression, changes in the structure of the skin or stress urinary incontinence in women. It has been documented that the risk of ischemic heart disease increases significantly after the onset of menopause which is reflected in the lowering of estrogen levels. These hormones are responsible for changes both in the lipid profile and in the vascular wall which significantly increases the likelihood of atherosclerotic plaque formation.

Hypertension is the most important cardiovascular risk factor affecting morbidity and mortality due to cardiovascular disease. It is estimated that there are as many as 34% of adult Poles. The incidence of hypertension increases with age in both women and men and significantly greater increases are observed in perimenopausal women.

An equally important and growing health and economic problem in Poland is heart failure. It is estimated that up to 700,000 patients in our country are struggling with this disease and the proportion of women in this group is constantly growing. This is the third reason for the death of women in Poland causing more deaths than cancer.

The influence of menopause on the occurrence of heart failure in a group of women with controlled hypertension remains unclear and is the subject of ongoing research. Similarly, there is still no convincing data on the increased risk of organ complications of arterial hypertension in the group of postmenopausal women.

Research carried out as part of this work will supplement the current knowledge on the impact of menopause in the population of women with hypertension on the risk of heart failure and complications of organ hypertension. Thanks to the observed relationships, it will be possible to early start the appropriate diagnostic procedure, the selection of personalized treatment and the development of a model of cardiac care for women in the perimenopausal period and thus, improve quality and extend their life.

Aim of the study: assessment of the influence of menopause on the ratios of myocardial efficiency, hemodynamic parameters and body composition in women aged > 40 years.

Detailed objectives:

* the influence of menopause on the body weight of the subjects assessed by the electrical bioimpedance method (BIA - BioelectricalImpedance Analysis)
* influence of menopause on early echocardiographic indices of heart failure and exercise capacity assessed objectively in spiroergometric study
* influence of menopause on endothelial function and central pressure assessed with the sphygmocor device (Atcor, Australia)
* influence of menopause on the concentration of biomarkers: asymmetric dimethylarginine (ADMA), NT-proBNP and neprilysin
* influence of menopause on the thickness of the intima-media complex

Methods:

* Subject and physical examination (BMI, waist measurement) and analysis of medical records
* Resting 12-lead electrocardiogram
* Transthoracic Echocardiography: a study will be performed on all patients using the GE Vivid E95 device according to current guidelines. The measurements of heart cavities, left ventricular volume and left ventricle ejection fraction calculated on the basis of Simpson's two-plane method will be evaluated. The mass of the left ventricle will be calculated using the Devereux formula. Evaluation of the left atrium with volume measurement will be performed. In addition, the assessment of cardiac output, mitral inflow with evaluation of the isovolumetric diastole time, speed of fast filling wave E, inflow wave velocity associated with left atrial contraction A, E / A ratio, rapid wave filling deceleration (E) of the mitral inflow, left atrial inflow with assessment of the maximal retrograde flow velocity in the lung veins, myocardial velocity in the study tissue Doppler technique with evaluation of the mitral ring velocity in the early stage of diastole E 'and late phase diastole A', systolic speed of the mitral annulus S ', E' / A 'ratio, E / E ratio and measurements of regional myocardial strain including global peak indices early and late diastolic deformities as well as echocardiographic vascular stiffness indexes.
* Biomarker Concentrations: blood taken from a vein by a vacuum (butterfly) system will be collected 10 ml of blood for the determination of selected biomarkers. Blood for the determination of biomarker concentration will be taken after inclusion into the study (the serum for determinations will be stored at -70 ° C and the assays will be performed using dedicated enzyme immunoassays after the first thawing of the samples, after collecting the entire pool.
* Body composition analysis using electrical bioimpedance (BIA). It is a method of analyzing fat, muscle and bones with the use of electricity. Particular tissues of the body contain a diversified amount of water, and therefore differ in the degree of electrical conduction. During the test, the amount of muscle, fat, visceral (abdominal) tissue, total water content in the body, bone mass, daily energy demand, metabolic age and, of course, body weight are measured. Methodology: the patient stands on a scale that contains electrodes. Then he sends weak current pulses to the organism (intensity 0.8-1mA, which is virtually imperceptible by human). The impedance or resistance of the body's tissues to the current is measured. A special computer program analyzes the individual bioelectrical impedance.
* Non-invasive assessment of haemodynamic parameters using the sphygmocor device (Atcor, Australia) with the assessment of vascular stiffness parameters such as: PWV (Pulse Wave Velocity), PWA (Pulse Wave Analysis), Alx (augmentation index) and central pressure
* Measurement of the intima-media complex All patients will be tested using the GE Vivid E95 device
* A spirometric stress test with the MetaLyzer 3B device is used to assess physical performance which translates into a clinical assessment of the patient's condition. The exercise test is carried out on a treadmill or a cycloergometer. During the effort, the respiratory gases are measured. One of the most important parameters being evaluated is the maximum oxygen consumption (VO2max). While in patients with cardiac diseases due to the difficulty in achieving their VO2max, the peak oxygen consumption (VO2 peak) is usually assessed. Other parameters assessed are: oxygen consumption (VO2), elimination of carbon dioxide (VCO2), oxygen consumption at the anaerobic threshold (VO2AT) and ventilation volume (VE). A spirometric stress test allows you to set an anaerobic threshold (AT). This is the intensity of the effort at which energy begins to be delivered as a result of anaerobic transitions. The anaerobic threshold can be determined by a non-invasive method using exhaust gas analysis. For this purpose, the V-slope method is used, in which the dependence of oxygen consumption (VO2) on the elimination of carbon dioxide (VCO2) is analyzed. The anaerobic threshold is the point at which the increase in VCO2 production exceeds the increase in O2 consumption.
* Statistical analysis. Statistical calculations will be made using statistical packages STATISTICA PL 10, SPSS 21, R-project 3.0.1 (packages: rms and predictAbel).

The Spearman rank correlation coefficients will be used to assess the dependencies between variables measured on an ordinal scale. Significant variables in the one-dimensional analysis (at the p <0.10 significance level) will be used to build multivariate logistic regression models. The quality of individual models and the usefulness of subsequent markers will be assessed using ROC curves [with the optimal cut-off points for which sensitivity, specificity and negative predictive power will be determined, also odds ratios OR with 95% confidence interval (95% CI) ], reclassification tables, NRI and IDI meters. Analysis of the endpoints will be performed using Kaplan-Meier curves.

ELIGIBILITY:
Inclusion Criteria:

About 100 women aged> 40 years will be included in the study with diagnosed pharmacologically controlled hypertension, including:

Group I-about 50 women > 40 years before the onset of menopause Group II - approximately 50 women > 1 year after the onset of menopause

Exclusion Criteria:

unstable hypertension;

* diagnosed heart failure or typical symptoms of heart failure;
* documented: hyperandrogenism, hyperendogenism, insulin resistance, premature ovarian failure, polycystic ovary syndrome;
* previous myocardial infarction;
* diagnosed cardiomyopathy (hypertrophic, dilated, restrictive, puerperal, tachyarrhythmic);
* storage diseases;
* stroke, TIA, an intracerebral bleeding;
* severe hyperthyroidism or hypothyroidism;
* pregnancy or lactation;
* chronic kidney disease in stage IV, V according to NKF and patients undergoing dialysis;
* documented cancer process;
* patient's inability to cooperate and / or give informed consent not to participate in a research;
* alcohol and drug abuse;
* active autoimmune disease;
* taking immunosuppressive, cytostatic drugs, glucocorticoids or antiretroviral drugs;
* bone marrow transplant or other organ transplantation, treatment with blood products during the last 6 months;
* active systemic infection;
* HBV, HCV or HIV infection or a positive result for the presence of HbS antigen or anti-HCV antibodies;
* surgery or serious injury in the last month;
* vaccination interview in the last 3 months;
* patients who have not expressed their informed consent to participate in the study

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Study Population: Women hospitalised in Department of Cardiology and Congenital Malformations of Adults Polish Mother's Memorial Hospital Research Institute
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
AMH | up to 2 years
  Anti-Müllerian Hormone

CONTACTS AND LOCATIONS:
Overall Officials: Agata Bielecka-Dąbrowa, MD PhD, Study Chair — Heart Failure Unit, Department of Cardiology and Congenital Malformations of Adults, Polish Mother's Memorial Hospital Research Institute
Locations (1):
- Heart Failure Unit, Department of Cardiology and Congenital Malformations of Adults, Polish Mother's Memorial Hospital Research Institute, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang N, Shao H, Chen Y, Xia F, Chi C, Li Q, Han B, Teng Y, Lu Y. Follicle-Stimulating Hormone, Its Association with Cardiometabolic Risk Factors, and 10-Year Risk of Cardiovascular Disease in Postmenopausal Women. J Am Heart Assoc. 2017 Aug 30;6(9):e005918. doi: 10.1161/JAHA.117.005918. PMID 28855169